CLINICAL TRIAL: NCT06878209
Title: Is Cough a Predisposing Factor for Hemorrhoids? A Prospective, Analytical Study
Brief Title: Cough and Hemorrhoids
Status: Recruiting | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Sabri Serhan OLCAY, Assistant Professor, Muğla Sıtkı Koçman University
Other Study IDs: 35
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-03

CONDITIONS: Hemorrhoid; Cough; Cough Duration; Cough Frequency; Cough Severity; Hemorrhoids, Internal
Keywords: cough, hemorrhoid
MeSH Terms: conditions — Hemorrhoids; Cough

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- coughing hemorrhoids: Patients diagnosed with hemorrhoidal disease in the general surgery outpatient clinic of our hospital

SUMMARY:
The aim of the study is to investigate the relationship between hemorrhoids and cough by assessing the symptoms, duration, and severity of cough in patients who will present to the general surgery outpatient clinic of Muğla Education and Research Hospital (MERH) with symptoms such as bleeding, pain, itching, fecal leakage, prolapse, and mucus discharge. These patients will be diagnosed with hemorrhoidal disease through rectal examination to detect anal pathology and will be graded according to mucosal prolapse. Our study will aim to determine whether cough is a predisposing factor for hemorrhoids by evaluating the presence, duration, and frequency of cough symptoms in patients with hemorrhoids. The study will be designed as a cross-sectional, analytical, and descriptive study. Between March 2025 and June 2025, patients with newly diagnosed hemorrhoids who will present to the MEAH General Surgery Outpatient Clinic will undergo physical examinations and will be assessed for cough symptoms. Evaluations will include height and weight measurements, the Leicester Cough Questionnaire, the Cough Visual Analog Scale (VAS) questionnaire, duration of cough (categorized as acute if shorter than 4 weeks, or chronic if longer than 4 weeks), timing of cough (day, night, or all day), comorbidities (such as COPD, asthma, chronic bronchitis, interstitial lung disease, idiopathic pulmonary fibrosis, and others), and smoking history (active, former, or never smoked). The primary endpoint will be to compare the relationship between the severity of hemorrhoids and the duration and frequency of cough in patients with both conditions. The secondary endpoint will be to compare the grade of hemorrhoids with comorbid chest diseases in these patients. The tertiary endpoint will be to compare the degree of hemorrhoids with the smoking history of patients who have both hemorrhoids and cough.

DETAILED DESCRIPTION:
Hemorrhoids are a collection of vascular tissue, smooth muscle, and connective tissue arranged in an inner column along the anal canal. Although they are normal structures, the term "hemorrhoids" refers to a pathological or symptomatic process. Internal hemorrhoids are located above the dentate line and are lined by columnar epithelium, which is innervated by visceral nerve fibers and not associated with pain, depending on the degree of prolapse, according to the Goligher classification. External hemorrhoids lie below the dentate line, are innervated by somatic nerves, and are usually asymptomatic.

Although the most common pathophysiologic cause of hemorrhoids is increased anal pressure at rest, the exact etiologic cause remains unclear. Factors that increase intra-abdominal pressure (IAP), such as straining during a bowel movement, prolonged sitting on the toilet, constipation/diarrhea, obesity, pregnancy, and age-related tissue weakening, can contribute to hemorrhoid development. However, the risk factors for hemorrhoids have not been sufficiently investigated.

The co-contraction of the thoracic, abdominal, and pelvic muscles results in a voluntary or reflex movement. This movement increases intrathoracic and intra-abdominal pressure (IAP), with IAP averaging 81.4-107.6 mmHg during coughing, compared to an average of 16.7 mmHg in the sitting position . The effect of coughing on IAP and its possible complications have been reported in case studies (e.g., urinary incontinence, pelvic organ prolapse) and electromyography studies.

A. Sadiqa et al. reported that hemorrhoids may develop as a gastrointestinal complication of coughing, but the relationship between cough and hemorrhoids has never been prospectively investigated.

Although there are no studies on the prevalence of hemorrhoids in our country, it is the third most common gastrointestinal diagnosis in the USA, with approximately 4 million outpatient and emergency department visits per year. The epidemiology of hemorrhoids has been theorized but remains largely unsupported by reliable research. Simply put, the commonly believed risk factors for hemorrhoids have not been adequately investigated. From an epidemiologic standpoint, whether coughing is a predisposing factor for hemorrhoids will be investigated for the first time in our study. We believe that this study may provide valuable insights for determining goals and strategies for the treatment and management of hemorrhoids, optimizing resource utilization, and offering evidence-based recommendations to patients. The study will be conducted using a prospective observational data collection method. The sample size was calculated using G*Power 3 software (Institute of Experimental Psychology, Heinrich Heine University, Germany). Power analysis showed a medium effect size (Cohen's d: 0.5), and the minimum number of samples required to detect a statistical difference at 95% power and a significance level of α = 0.05 was 134.

Patients diagnosed with hemorrhoidal disease in the general surgery outpatient clinic of our hospital will be included in the study. Demographic information, such as age, gender, educational status, and occupational status, will be recorded for patients who sign the voluntary informed consent form. Additionally, data on the duration of hemorrhoidal disease based on symptomatology, the stage of the disease according to the Goligher classification, the presence of additional proctologic diseases, the presence or absence of constipation symptoms, the severity of bleeding, nutrition and toilet habits, and previous medical or surgical treatments for hemorrhoidal disease will be collected.

Information regarding the presence of cough, additional obstructive pulmonary diseases, medications, smoking or alcohol use, the Leicester Cough Questionnaire, and the Cough Visual Analog Scale (Cough VAS) will also be recorded. Patients with cough will be referred to the Department of Chest Diseases for diagnostic and therapeutic evaluation to investigate the etiology of cough.

If sufficient information is collected from a sufficient number of patients who meet the study criteria, the data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Being 18 years of age or older
2. Speaking and understanding Turkish
3. To be mentally and cognitively capable of understanding the questions asked
4. To agree to participate in the research
5. individuals diagnosed with hemorrhoidal disease

Exclusion Criteria:

1. Those with existing proctologic disease other than hemorrhoidal disease and pelvic floor disease
2. Patients with previous surgery for hemorrhoidal disease
3. Patients with hemorrhoidal disease caused by portal hypertension
4. Patients during pregnancy and diagnosed with postpartum hemorrhoidal disease
5. those with benign prostatic hyperplasia or neurogenic bladder that may cause increased intra-abdominal pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with hemorrhoidal disease in MERH General Surgery Outpatient Clinic who meet the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-09-14 (Estimated); Study Completion 2025-10-14 (Estimated)

PRIMARY OUTCOMES:
Leicester cough questionnaire | day 1
  The primary endpoint is to compare the relationship between the severity of hemorrhoids and the duration and frequency of cough in patients with hemorrhoids and cough.

SECONDARY OUTCOMES:
Comobidities | day 1
  The secondary endpoint was to compare the grade of hemorrhoids and comorbidities of chest diseases in patients with hemorrhoids and cough.

OTHER OUTCOMES:
Smoking | day 1
  Comparison of the degree of hemorrhoids and smoking history of patients with hemorrhoids and cough is the tertiary endpoint.

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Training and Research Hospital, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided